CLINICAL TRIAL: NCT02336555
Title: A Randomized Clinical Trial to Study the Efficacy, Safety, and Tolerability of MK-8291 in Subjects With Post-Herpetic Neuralgia With Allodynia
Brief Title: The Efficacy of MK-8291 in Participants With Post-herpetic Neuralgia (PHN) With Allodynia (MK-8291-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8291-012; 2014-002396-28 (EudraCT Number); MK-8291-012 (Other: Merck)
Record Dates: First submitted 2015-01-05; First posted 2015-01-13 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-8291 → Placebo (Experimental): In Treatment Period 1, participants were orally administered 10 mg MK-8291 once daily on Days 1 and 2, twice daily on Days 3 to 27, and once daily on Day 28 of the period. After Treatment Period 1, participants were to undergo a minimum of a 7-day Washout Period, which was followed by Treatment Period 2. In Treatment Period 2, participants were orally administered Placebo once daily on Days 1 and 2, twice daily on Days 3 to 27, and once daily on Day 28 of the period. (Total duration of treatment: up to approximately 63 days)
  Interventions: Drug: MK-8291; Drug: Placebo
- Placebo → MK-8291 (Experimental): In Treatment Period 1, participants were orally administered Placebo once daily on Days 1 and 2, twice daily on Days 3 to 27, and once daily on Day 28 of the period. After Treatment Period 1, participants were to undergo a minimum of a 7-day Washout Period, which was followed by Treatment Period 2. In Treatment Period 2, participants were orally administered 10 mg MK-8291 once daily on Days 1 and 2, twice daily on Days 3 to 27, and once daily on Day 28 of the period. (Total duration of treatment: up to approximately 63 days)
  Interventions: Drug: MK-8291; Drug: Placebo

INTERVENTIONS:
Drug: MK-8291 — MK-8291 oral tablets
Drug: Placebo — Placebo oral tablets

SUMMARY:
This study aims to determine whether MK-8291 is effective in reducing pain in participants with post-herpetic neuralgia (PHN) with allodynia.

The primary hypothesis is that when compared to placebo, treatment with MK-8291 reduces the change from Baseline in participant-reported pain intensity by 1 on an 11-point numeric rating scale.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant female (and/or partner) agrees to use two acceptable methods of birth control throughout the trial until 2 weeks after the last dose of treatment
* female is postmenopausal or surgically sterile
* has a clinical diagnosis of PHN with allodynia for at least 3 months duration after healing of rash
* has a body mass index (BMI) =< 35 kg/m^2, inclusive
* is in good health, with exception of PHN
* is on a stable dose for at least 30 days prior to screening if taking any of the following: opioids, non-opioids, paracetomol, non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, antidepressants
* is a nonsmoker or has not used nicotine or nicotine containing products for at least prior 3 months

Exclusion Criteria:

* has a non-PHN chronic pain state
* has a history of clinically significant and inadequately treated endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* has a history of malignant cancer
* has a history or presence of esophagitis
* has a history of significant multiple and/or severe allergies (e.g. food, drug, latex), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* is positive for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV)
* had major surgery, donated or lost approximately 500 mL of blood within 4 weeks prior to screening
* has participated in another investigational trial within 4 weeks prior to screening
* has a history of risk factors for Torsades de Pointes, has hypokalemia or hypomagnesemia
* has a history or presence of clinically significant cardiac arrhythmia, taking substances with the target of reducing heart rate and or exercising endurance sports
* has had an injection of local anesthetics or steroids in the region affected by PHN, within 35 days prior to randomization
* anticipates using prescription and non-prescription drugs or herbal remedies during trial
* consumes excessive amounts of alcoholic or caffeinated beverages
* uses cannabis, any illicit drugs, or has a history of drug (including alcohol) abuse within 12 months of screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males and females with post-herpetic neuralgia (PHN) with allodynia, at least 18 years of age (inclusive) were enrolled in this study.
Period: Treatment Period 1 (28 Days)
Arm/Group | MK-8291 → Placebo | Placebo → MK-8291
Started | 18 | 17
Completed | 16 | 16
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 2 | 0
Period: Treatment Period 2 (28 Days)
Arm/Group | MK-8291 → Placebo | Placebo → MK-8291
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8291 → Placebo | Placebo → MK-8291 | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (16.7) | 54.7 (13.5) | 55.7 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Numerical Rating Scale (NRS) Pain Intesity Score at Baseline [Mean (Standard Deviation); unit: Score on a scale] — Participants completed a pain intensity questionnaire, the Numerical Rating Scale (NRS), in the morning prior to taking study treatment at Baseline (Day 1) in each treatment period. The NRS assessed the intensity of Post-herpetic Neuralgia (PHN) pain during the preceding 24-hour period on an 11-point numeric rating scale (range: 0=no pain to 10=pain as bad as you can imagine), with a higher score indicating worse pain levels. The mean pain intensity score at Baseline is presented by treatment sequence. Population: Two MK-8291→Placebo and one Placebo→MK-8291 participants did not have Baseline NRS Pain Intensity Scale scores.
  Score on a scale
    number analyzed (Participants) | 16 | 16 | 32
    (all) | 6.63 (1.02) | 6.00 (0.97) | 6.31 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Intensity at Week 4 of Each Treatment Period
Description: Participants completed a pain intensity questionnaire, the Numerical Rating Scale (NRS), in the morning prior to taking study treatment at Baseline (Day 1) in each treatment period, and then daily up to Day 28 in each treatment period. The NRS assesses the intensity of Post-herpetic Neuralgia (PHN) pain during the preceding 24-hour period on an 11-point numeric rating scale (range: 0=no pain to 10=pain as bad as you can imagine). The mean score in pain intensity of Week 4 (Days 22 to 28) minus the mean score at Baseline is presented, with a negative change representing improvement (or reduction) in pain intensity. In comparison to placebo, a reduction (difference in the change from Baseline) of 1 on the 11-point NRS is expected.
Time Frame: Baseline and Days 22-28 of each treatment period (Up to approximately 63 days)
Population: The population consisted of participants who complied with the protocol sufficiently to ensure that these data would be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- MK-8291: Participants were orally administered 10 mg MK-8291 once daily on Days 1 and 2, twice daily on Days 3 to 27, and once daily on Day 28 of a treatment period. (Up to 28 days in each treatment period)
- Placebo: Participants were orally administered Placebo once daily on Days 1 and 2, twice daily on Days 3 to 27, and once daily on Day 28 of a treatment period. (Up to 28 days in each treatment period)
Arm/Group | MK-8291 | Placebo
Number analyzed (Participants) | 30 | 32
Score on a scale | -1.776 [-2.442 to -1.110] | -1.263 [-1.742 to -0.785]
Statistical Analysis 1: Comparison: MK-8291 vs Placebo; Test type: Superiority; p = 0.075, Linear mixed model — Linear mixed model with a posterior probability evaluation for the treatment effect; One-sided p-value and a posterior probability greater than 90% that the treatment effect is less than 0; Mean Difference (Final Values) = -0.452, 95% CI 2-sided [-1.076 to 0.172]

2. Secondary Outcome: Percentage of Participants Achieving a 30 Percent or Greater Change From Baseline to Day 28 in Pain Intensity
Description: Participants completed a pain intensity questionnaire, the Numerical Rating Scale (NRS) in the morning before taking study treatment at Baseline (Day 1) in each treatment period, and then daily from Day 1 up to Day 28 in each treatment period. The NRS assesses the intensity of PHN pain during the preceding 24-hour period on an 11-point numeric rating scale (range: 0=no pain to 10=pain as bad as you can imagine). This was a binary outcome denoting whether the participant reported a percent change from Baseline to Week 4 (Days 22 to 28) in the mean pain intensity score greater than 30%. The percentage of participants who reported a 30% or greater change from Baseline to Day 28 of each treatment period is presented.
Time Frame: Baseline and Day 28 in each treatment period (Up to approximately 63 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-8291 | Placebo
Number analyzed (Participants) | 30 | 32
Percentage of participants | 36.7 [19.9 to 56.1] | 34.4 [18.6 to 53.2]
Statistical Analysis 1: Comparison: MK-8291 vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.073, 95% CI 2-sided [0.446 to 2.580] — Logistic regression model with factors for treatment & baseline pain intensity

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 14 days after last dose of study treatment (Up to a total of approximately 80 days)
Description: All-Cause Mortality Population: All randomized participants. Adverse Events Population: All participants who received at least one dose of study treatment.
Arm/Group | MK-8291 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/33
Other Adverse Events (participants affected / at risk) | 21/34 | 6/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8291 (N=34) | Placebo (N=33)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8291 (N=34) | Placebo (N=33)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
PHOTOPSIA (Eye disorders) | 7 (7) | 0 (0)
VISION BLURRED (Eye disorders) | 3 (5) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (10) | 1 (1)
VOMITING (Gastrointestinal disorders) | 5 (8) | 0 (0)
ASTHENIA (General disorders) | 3 (4) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PERIODONTITIS (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BALANCE DISORDER (Nervous system disorders) | 3 (3) | 1 (1)
BURNING SENSATION (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 13 (25) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (3) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 2 (2) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.